CLINICAL TRIAL: NCT05206591
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled, Multicenter Phase III Study to Investigate the Efficacy and Safety of Secukinumab (Cosentyx®) 300 mg Administered Subcutaneously in Patients With Active Peripheral Spondyloarthritis (pSpA).
Brief Title: Study to Demonstrate the Efficacy and Safety of Secukinumab up to 224 Weeks in Subjects With Active Peripheral Spondyloarthritis (pSpA).
Acronym: CAIN457X12301
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial terminated due to strategic decision of senior management
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457X12301
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Active Peripheral Spondyloarthritis (pSpA)
Keywords: secukinumab, active peripheral spondyloarthritis (pSpA)
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Secukinumab 300 mg s.c
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Placebo s.c.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Secukinumab — Secukinumab 300 s.c.
  Arms: Secukinumab
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of subcutaneous (s.c) secukinumab in comparison with placebo for participants with two subtypes of active pSpA i.e. undifferentiated pSpA and chronic reactive arthritis, and with an inadequate response to conventional therapy despite current or previous Non-steroidal Anti Inflammatory Drugs (NSAIDs) and/or csDMARDs. Additionally, the study aims to evaluate efficacy and safety of continuing versus withdrawing secukinumab therapy in maintaining remission in the study population.

DETAILED DESCRIPTION:
This is a randomized, parallel-group, double-blind, placebo-controlled, multicenter, Phase III study designed to assess efficacy and safety of secukinumab compared to placebo in adult patients with active pSpA, composed of the subsets of undifferentiated pSpA and chronic reactive arthritis. Approximately 324 eligible participants with pSpA will enroll into the study with approximately 162 participants in each of the double-blind arms. This population will be comprised of approximately 292 participants with undifferentiated pSpA and approximately 32 participants with chronic reactive arthritis.

The participants will be stratified 1:1 ratio at randomization (Baseline) according to:

* High Sensitivity C-reactive Protein (hsCRP) level: Participants will be equally stratified based on hsCRP (≤5mg/L) or hsCRP (>5 mg/L) as measured at Screening Visit 2 (SV2) with the hsCRP (≤5mg/L) strata capped at 50%.
* Sub-type of pSpA: Approximately 90% of randomized participants will be diagnosed with undifferentiated pSpA and up to 10% participants with chronic reactive arthritis.

The trial consists of 5 periods: a screening, double-blind treatment, randomized withdrawal, an open label treatment and safety follow-up period, detailed below:

1. Screening period- Up to 8 weeks to assess participant's eligibility, composed of 2 visits - SV1 and SV2.
2. Double-blind Treatment period - Baseline (BSL) (Week 0) to Week 56 [Treatment Period 1]

   Eligible participants will be randomized at BSL (Week 0) in a 1:1 ratio to one of the following double-blind arms:
   * Arm 1 (N=162 participants): Secukinumab 300 mg s.c. at Week 0, 1, 2, 3, 4, then every 4 weeks thereafter up to and including Week 52.
   * Arm 2 (N= 162 participants): Placebo s.c. at Week 0, 1, 2, 3, 4, then every 4 weeks thereafter up to and including Week 52.
3. Randomized Withdrawal- (Week 56 to Week 108) [Treatment Period 2]
4. Open-label Treatment period- (Week 20 to Week 216) [Treatment Period 3]
5. Safety Follow-up period - Following the EOT visit at Week 216, there will be an End of Treatment (EOS) visit at Week 224 for safety assessments

The primary endpoint analysis will be performed after all participants have completed the Week 16 visit. The investigators, site personnel and monitors will continue to remain blinded to the original treatment assignment that each participant received at randomization until after the database lock for final analysis.

Analysis Plan A is planned after participants have completed the Week 16 assessments. Analysis Plan B is planned after participants have completed the Week 52 assessments in order to support regulatory submission and/or publication purposes. The analysis at Week 108 will be conducted after all participants complete the Treatment Period 2. The final analysis will be conducted after all participants complete the study. Additional analyses may be performed to support interactions with health authorities, as necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Participant must be able to understand and communicate with the investigator and comply with the requirements of the study.
3. Male or non-pregnant, non-lactating female participants at least 18 years of age.
4. Participant meets ASAS criteria for classification of pSpA:

   * Participant must have current arthritis (asymmetric or predominantly in the lower limbs) or enthesitis (except for enthesitis only along the spine
   * , sacroiliac joints and/or chest wall) or dactylitis. AND at least one of the following SpA features:
   * Anterior uveitis in past confirmed by a qualified medical professional (participants with current ongoing uveitis are excluded from participation in the study)
   * Evidence of preceding infection (acute diarrhea or non-gonococcal urethritis or cervicitis 1 month before arthritis)
   * HLA-B27 positivity
   * Sacroiliitis on imaging; based on prior magnetic resonance imaging (MRI) or X-ray OR at least 2 of the following SpA features:
   * Arthritis (past or present diagnosis), adequately documented and identified, or diagnosed by a qualified medical professional
   * Enthesitis (any location, past or present diagnosis), adequately documented and identified, or diagnosed by a qualified medical professional
   * Dactylitis (past or present diagnosis) adequately documented and identified, or diagnosed by a qualified medical professional
   * Inflammatory back pain (past or present) Note: If there is concurrent inflammatory back pain it must be < 2 on NRS score for total back pain & nocturnal back pain (score 0-10) and the peripheral symptomatology of pSpA must be the predominant symptoms at study entry, based on the investigator's judgment at baseline.
   * Family history for SpA.
5. Diagnosis of pSpA with evidence of active disease as manifested by

   * Patient's global assessment of disease activity (0-100 VAS) ≥ 40 mm, and
   * Patient's global assessment of pain (0-100 VAS) ≥ 40 mm, and
   * At least one of the following:
   * ≥ 2 joints that are both tender and swollen
   * ≥ 2 sites of severe enthesitis as assessed by the investigator and ≥ 1 joint that is both tender and swollen
   * ≥ 2 digits with dactylitis and ≥1 joint that is both tender and swollen not associated with dactylitis
6. Rheumatoid Factor (RF) and Anti-cyclic citrullinated peptides (anti-CCP) antibodies negative at screening.
7. Duration of symptoms of at least 6 months.
8. Participant should have been on at least 2 different non-steroidal anti-inflammatory drugs (NSAIDs) at the highest recommended dose for at least 4 weeks in total prior to randomization with an inadequate response or failure to respond, or less if therapy had to be withdrawn due to intolerance, toxicity or contraindications.
9. Participant taking methotrexate (≤ 25 mg/week), or sulfasalazine (≤ 3 g/day), or hydroxychloroquine (≤ 400 mg/day) are allowed to continue their medication and must have taken it for at least 3 months and must be on a stable dose and route of administration for at least 4 weeks prior to randomization. Only one of these csDMARDs can be continued during the study.
10. Participant on stable MTX must be on folic acid supplementation at randomization. 11.Participant taking systemic corticosteroids must be on a stable dose of ≤ 10 mg/day prednisone or equivalent for at least 2 weeks before randomization.

Exclusion Criteria:

1. Current or previous diagnosis of :

   * Psoriasis (PsO) and/or nail changes consistent with PsO diagnosed by a qualified medical professional
   * PsA diagnosed by a qualified medical professional
   * Inflammatory bowel disease (IBD) diagnosed by a qualified medical professional
   * axSpA (AS or nr-axSpA) diagnosed by a qualified medical professional
2. Meets ASAS axSpA criteria as manifested by ALL of:

   a. Inflammatory back pain for at least 3 months b. Onset before 45 years of age c.

   Sacroiliitis on MRI with ≥ 1 SpA feature OR HLA-B-27 positive with ≥2 SpA features
3. Score of ≥2 on numerical rating scale (NRS)-score for total back pain and nocturnal back pain (score 0-10)
4. History of a confirmed diagnosis of any inflammatory joint disorder other than pSpA (e.g., rheumatoid arthritis, gouty arthritis, other crystalline arthritis, systemic lupus erythematosus, or any arthritis with onset prior to age 16 years such as juvenile idiopathic arthritis).
5. Prior exposure to TNF-i's or other biologic immunomodulating agents, investigational or approved
6. Active ongoing inflammatory diseases other than pSpA that might confound the evaluation of the benefit of secukinumab therapy (e.g., uveitis).
7. Current or previous diagnosis of fibromyalgia by a qualified medical professional
8. Diagnosis of synovitis associated with primary osteoarthritis
9. Diagnosis of septic arthritis, sarcoidosis, seronegative RA, or erosive osteoarthritis
10. Current severe progressive or uncontrolled disease, which in the judgment of the clinical investigator renders the particpant unsuitable for the trial.
11. History of clinically significant liver disease or liver injury indicated by abnormal liver function tests, such as SGOT (AST), SGPT/ Alanine transaminase (ALT), Alkaline

    phosphatase (ALP) and serum bilirubin. The investigator should be guided by the following criteria:
    * Any single parameter may not exceed 2 x the upper limit of normal (ULN). A single parameter elevated up to and including 2 x ULN should be re-checked once more as soon as possible, and in all cases, at least prior to randomization, to rule-out laboratory error.
    * If the total bilirubin concentration is increased above 2 x ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum bilirubin should not exceed the value of 1.6 mg/dL (27 µmol/L).
12. Screening total White Blood Cells (WBC) count <3,000/μl, or platelets <100,000/μl or neutrophils <1,500/μl or hemoglobin <8.5 g/dl (85 g/L).
13. Plans for administration of live vaccines during the study period or 6 weeks prior to randomization.
14. Significant medical problems or diseases, including but not limited to the following: uncontrolled hypertension (≥160/95 mmHg), congestive heart failure (New York Heart Association status of class III or IV), uncontrolled diabetes, or very poor functional status precluding ability to perform self-care.
15. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human Chorionic Gonadotropin (hCG) laboratory test.
16. History or evidence of ongoing alcohol or drug abuse, within the last six months before randomization.
17. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment. Effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post- ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant
    * Barrier methods of contraception: Condom or Occlusive cap (e.g. diaphragm or cervical/vault caps)
    * Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS).

    In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    NOTE:

    Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms). Women are considered not of child bearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

    If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.
18. Previous treatment with any cell-depleting therapies including but not limited to anti- CD20 or investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti- CD19).
19. Use of other investigational drugs at the time of enrollment, or within 5 half- lives of enrollment, or within 4 weeks until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations.
20. Use or planned use of prohibited concomitant medication (see Section 6.2.2).
21. History of lymphoproliferative disease or any known malignancy, or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for skin Bowen's disease, or basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non- invasive malignant colon polyps that have been removed).
22. Presence of significant medical problems which in the opinion of the investigator will interfere with study participation, including but not limited to the following: participants with severely reduced kidney function (estimated glomerular filtration rate (eGFR) <29 ml/min/1.73m2).
23. History of hypersensitivity to any of the study drug constituents.
24. Any medical or psychiatric condition, which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.
25. Chest X-ray or MRI (at Screening Visit 1) with evidence of ongoing infectious or malignant process obtained within 3 months of screening and evaluated by a qualified physician.
26. Active systemic infection during the last two weeks (exception: common cold) prior to randomization or any infection that reoccurs on a regular basis.
27. Underlying conditions (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the participant and/or places the participant at unacceptable risk for receiving an immunomodulatory therapy
28. Known infection with Human Immunodeficiency Virus (HIV), hepatitis B or hepatitis C at screening or randomization.
29. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test as indicated in the assessment schedule. Participants with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the participant has no evidence of active tuberculosis. After active tuberculosis has been excluded, treatment for latent tuberculosis according to local country guidelines must have been initiated prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-16 (Estimated); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-06-12 (Estimated)

PRIMARY OUTCOMES:
Modified Peripheral SpondyloArthritis Response Criteria (mPSpARC) | Week 16
  To demonstrate the superiority of secukinumab compared to placebo based on Modified Peripheral SpondyloArthritis Response Criteria mPSpARC40